CLINICAL TRIAL: NCT02304120
Title: Effects of a Sensorimotor Training on Postural Control and Pain: A Parallel, Single-blinded Randomised Controlled Trial
Brief Title: Sensorimotor Training in Low-back Pain Rehabilitation
Acronym: SeMoPoP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michael A. McCaskey (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor-Investigator, Michael A. McCaskey, Master of Science in Human Movement Science, Reha Rheinfelden
Organization: Reha Rheinfelden (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014-0873
Record Dates: First submitted 2014-11-17; First posted 2014-12-01 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Low Back Pain
Keywords: proprioception; postural control; sensorimotor training; uncontrolled manifold
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sensorimotor (Experimental): The experimental group will receive added PPT to the conventional physiotherapy. PPT will be applied by means of a neuro-orthopaedic medical device ("Posturomed®", see section 3.2). The "Posturomed" allows adaptive oscillation in the horizontal plane. Therapy instructions advise seven stages of difficulty. In all stages the patient is asked to provoke oscillation by stepping on site. After three steps, the patient must stand still on one leg for 2 seconds before he or she repeats the steps. Difficulty is increased by a) decreasing the damping through release of the breaks and b) through added juggling of a ball during the motor task (dual-task and divided attention). The next stage is reached once stabilisation in the previous stage is secured.
  Interventions: Other: Proprioceptive postural training; Other: Conventional physiotherapy
- Low-intensity activity (Active Comparator): Added to conventional therapy, as administered to all participants, the control group will do added treadmill walking. The control intervention will consist of 10 minutes of walking at comfortable pace. The patient will be instructed in treadmill functions and asked to set the speed between 2 and 4 km/h. The speed should be adjusted to the level where the patient would still be able to talk comfortably.
  Interventions: Other: Treadmill training; Other: Conventional physiotherapy

INTERVENTIONS:
Other: Proprioceptive postural training
  Other Names: Sensorimotor training
  Arms: Sensorimotor
Other: Treadmill training
  Arms: Low-intensity activity
Other: Conventional physiotherapy — All participating patients will attend usual care according to their treatment plan (taking part in the study does not affect the treatment plan). A physiotherapy referral requests 9 treatments, each of which takes 30 minutes. These will take place twice a week for 4.5 weeks. The study protocol does not dictate the content of the physiotherapy sessions themselves, but detailed documentation of provided treatments is required (therapy documentation sheet). Additionally, the aim of the physiotherapy sessions should always include reduction of muscular imbalances and optimisation of posture.

SUMMARY:
This study evaluates the effects of additional sensorimotor training (proprioceptive postural training, PPT) to conventional therapy in the treatment of chronic low-back pain. Half of the participants will receive instructed treadmill training as an active comparator against PPT. All participants receive conventional physiotherapy as prescribed by their treating medical doctors. It is expected that the PPT group will improve in postural control, proprioceptive, as well as pain and function outcomes to a significantly greater extent than the active control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with musculoskeletal low back pain (non-specific low back pain)
* Age ≥ 18 years

Exclusion Criteria:

* Known or suspected neurological diseases or lesions
* Traumatic injury of musculoskeletal system (fractures, tumours)
* Spinal pathologies (e.g., tumour, infection, fracture, and inflammatory disease)
* Previous spinal surgery
* Presence of any contraindication to exercise (fracture or cardiovascular limitations)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-12; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change of self-reported pain on 100mm Visual Analogue Scale (VAS) | Baseline (-4 days); Pre-Test (0 days); Post-Test (+25 days) and follow-up (+45 days)
Change of functional status recorded with the Oswestry Disability Index (ODI) | Baseline (-4 days); Pre-Test (0 days); Post-Test (+25 days) and follow-up (+45 days)

SECONDARY OUTCOMES:
Centre of Pressure | Baseline (-4 days); Pre-Test (0 days); Post-Test (+25 days) and follow-up (+45 days)
  Area of surface a the 95% confidence ellipse of centre of pressure displacement during postural task
Joint Repositioning Error (segmental) | Baseline (-4 days); Pre-Test (0 days); Post-Test (+25 days) and follow-up (+45 days)
  Repositioning acuity after surface perturbation.
Uncontrolled Manifold Index (UCM) | Baseline (-4 days); Pre-Test (0 days); Post-Test (+25 days) and follow-up (+45 days)
  Segmental joint configuration.

CONTACTS AND LOCATIONS:
Overall Officials: Michael A McCaskey, MSc, Principal Investigator — Reha Rheinfelden; Eling D. de Bruin, PD PhD, Study Chair — ETH Zurich; Corina Schuster-Amft, PT PhD, Study Chair — Reha Rheinfelden
Locations (1):
- Reha Rheinfelden, Rheinfelden, Canton of Aargau, Switzerland

REFERENCES:
- [Background] Scholz JP, Schoner G. The uncontrolled manifold concept: identifying control variables for a functional task. Exp Brain Res. 1999 Jun;126(3):289-306. doi: 10.1007/s002210050738. PMID 10382616
- [Derived] McCaskey MA, Wirth B, Schuster-Amft C, de Bruin ED. Postural sensorimotor training versus sham exercise in physiotherapy of patients with chronic non-specific low back pain: An exploratory randomised controlled trial. PLoS One. 2018 Mar 9;13(3):e0193358. doi: 10.1371/journal.pone.0193358. eCollection 2018. PMID 29522571
- [Derived] McCaskey MA, Schuster-Amft C, Wirth B, de Bruin ED. Effects of postural specific sensorimotor training in patients with chronic low back pain: study protocol for randomised controlled trial. Trials. 2015 Dec 15;16:571. doi: 10.1186/s13063-015-1104-4. PMID 26666457